CLINICAL TRIAL: NCT05360160
Title: A Phase I-II Study Investigating the All Oral Combination of the Menin Inhibitor SNDX-5613 With Decitabine/Cedazuridine (ASTX727) and Venetoclax in Acute Myeloid Leukemia (SAVE)
Brief Title: A Phase I-II Study Investigating the All-Oral Combination of the Menin Inhibitor SNDX-5613 With Decitabine/Cedazuridine (ASTX727) and Venetoclax in Acute Myeloid Leukemia (SAVE)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry); Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1059; NCI-2022-03312 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-04-13; First posted 2022-05-04 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SNDX-5613 (Experimental): Capsules by mouth 2 times every day (about 12 hours apart).
  Interventions: Drug: SNDX-5613
- Venetoclax (Experimental): Tablets by mouth on Days 1-14 of each cycle.
  Interventions: Drug: Venetoclax
- ASTX727 (Experimental): Tablets by mouth on Days 1-5 of each cycle.
  Interventions: Drug: ASTX727

INTERVENTIONS:
Drug: SNDX-5613 — Given by PO
  Arms: SNDX-5613
Drug: Venetoclax — Given by PO
  Arms: Venetoclax
Drug: ASTX727 — Given by PO
  Arms: ASTX727

SUMMARY:
Part 1b of this clinical research study is to find the highest tolerable dose of SNDX-5613 that can be given in combination with ASTX727 (a combination of the drugs decitabine/cedazuridine) and venetoclax for patients with acute myeloid leukemia (AML) or those with a mixed phenotype acute leukemia with a myeloid phenotype (MPAL).

Part 2 of this study is to learn if the dose of study drugs found in Part 1b can help to control AML/MPAL

DETAILED DESCRIPTION:
Primary Objectives:

Phase Ib

• To determine the safety, tolerability and recommended phase II dose (RP2D) of SNDX-5613 in combination with oral decitabine/cedazuridine (ASTX727) and venetoclax for patients with acute myeloid leukemia (AML).

Phase II

• To assess the efficacy of SNDX-5613 in combination with ASTX727 and venetoclax for patients with AML.

Secondary Objectives

• To assess overall survival, event-free survival and duration of response.

Exploratory Objectives

• To evaluate molecular and cellular markers that may be predictive of antitumor activity and/or resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 12 years with weight ≥ 40Kg.
2. ECOG performance status of ≤ 2.
3. Newly diagnosed (frontline cohort), who are not eligible for high-intensity induction chemotherapy or relapsed/refractory (R/R cohort) AML or myeloid phenotype MPAL with either KMT2Ar, or NUP98r, or NPM1c.
4. WBC must be below 25,000/ μL at time of enrollment. Patients may receive cytoreduction prior to enrollment.
5. Baseline ejection fraction must be > 40%.
6. Adequate hepatic function (direct bilirubin < 2x upper limit of normal (ULN) unless increase is due to Gilbert's disease or leukemic involvement, and AST and/or ALT < 3x ULN unless considered due to leukemic involvement, in which case direct bilirubin or AST and/or ALT < 5x ULN will be considered eligible).
7. Adequate renal function (creatinine clearance ≥ 30 mL/min) unless related to disease.
8. Willing and able to provide informed consent.
9. In the absence of rapidly proliferative disease, the interval from prior treatment to time of initiation will be at least 14 days for cytotoxic or non-cytotoxic (immunotherapy agent(s), or an interval of 5 half-lives of the prior therapy. Oral hydroxyurea and/or cytarabine (up to 2 g/m2) for patients with rapidly proliferative disease is allowed before the start of study therapy, as needed, for clinical benefit and after discussion with the PI. Concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted.
10. Women of childbearing potential must agree to adequate methods of contraception during the study and at least 3 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study and at least 3 months after the last treatment.

Exclusion Criteria:

1. Prior treatment with a menin inhibitor.
2. Patients with any concurrent uncontrolled medical condition, laboratory abnormality, or psychiatric illness which could place the patient at unacceptable risk of study treatment.
3. The use of other chemotherapeutic agents or anti-leukemic agents is not permitted during study with the following exceptions (1) intrathecal chemotherapy for prophylactic use or for controlled CNS leukemia. (2) use of hydroxyurea for patients with rapidly proliferative disease or for control of counts during differentiation syndrome. (3) use of steroids for treatment of differentiation syndrome.
4. Patients with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications.
5. Patients with a concurrent active malignancy under treatment.
6. Known active hepatitis B (HBV) or Hepatitis C (HCV) infection or known HIV infection.
7. Female subjects who are pregnant or breast-feeding.
8. Patient has an active uncontrolled infection.
9. Any of the following within the 6 months prior to study entry: myocardial infarction, uncontrolled/unstable angina, congestive heart failure (New York Heart Association Classification Class ≥II), life-threatening, uncontrolled arrhythmia, cerebrovascular accident, or transient ischemic attack.
10. QTc >470 msec using the Fridericia Formula.
11. History of a complete bundle branch block or high-degree atrioventricular block.
12. History of or any concurrent condition, therapy, or laboratory abnormality that in the Investigator's opinion might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate.
13. Clinically active central nervous system (CNS) leukemia.
14. Patients on immunosuppressive therapy post-HSCT at the time of screening with R/R leukemia (must be off all systemic immunosuppression therapy for at least 2 weeks and calcineurin inhibitors for at least 4 weeks). The use of topical steroids for cutaneous graftversus- host disease (GVHD) or stable systemic steroid doses less than or equal to 20 mg of prednisone daily are permitted.
15. Patients with Grade > 2 active acute GVHD, moderate or severe limited chronic GVHD, or extensive chronic GVHD of any severity.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
To establish the recommended phase II dose (RP2D) of SNDX-5613 in combination with oral decitabine/cedazuridine (ASTX727) and venetoclax for patients with acute myeloid leukemia (AML). | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ghayas Issa, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Garcia MB, Wang B, Sheikh I, El Hajjar G, McCall D, Nunez C, Gibson A, Lorenzi PL, Issa GC, Cuglievan B, Abbas HA. High-throughput proteomic profiling to evaluate differentiation syndrome with menin inhibition. Mol Cell Proteomics. 2026 Jan 30:101522. doi: 10.1016/j.mcpro.2026.101522. Online ahead of print. PMID 41621809
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT05360160/ICF_000.pdf